CLINICAL TRIAL: NCT04756479
Title: Predictors of Intrahospital Mortality in Older Patients Admitted Due to COVID-19 in the COVID-19 AGEBRU Study
Brief Title: Mortality Due to COVID-19 in the COVID-AGEBRU Study
Acronym: COVID-AGEBRU
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Murielle Surquin, Geriatrics Department, Brugmann University Hospital
Other Study IDs: COVID-19 AGE-BRUGMANN 2020/111
Record Dates: First submitted 2021-02-08; First posted 2021-02-16 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Covid19; Old Age; Debility; Morbidity, Multiple
MeSH Terms: conditions — COVID-19; Frailty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The COVID-Age Brugmann study aims to identify the clinical predictors of mortality risk in older patients admitted to an acute care unit due to COVID-19

DETAILED DESCRIPTION:
The COVID-19 disease has been shown to be associated to higher mortality risk and health adverse consequences. Despite of the fact that the SAR-COV2 virus has been shown that affects every populations, the negative impact is higher in older people, pointing this population as the most severely affected.

The COVID-Age Brugmann study aims to identify if comorbidity, geriatric syndromes, and health issues at admission are associated to mortality risk in older patients admitted to an acute care unit due to COVID-19

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 70 and older
* Patients admitted to an acute care geriatric unit due to COVID-19
* Patients with COVID-19 by PCR, serology or CT scan suggestive of this disease

Exclusion Criteria:

* No other demographic or clinical exclusion criteria will be applied

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Consecutive patients aged 70 and over hospitalized in an acute care unit in Brugmann university hospital, in Belgium, due to COVID-19 in the period Mars to June 2020.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
All-cause mortality during hospital admission (admission up to discharge time) | Through study completion, an average of one month.
  Vital status was obtained from medical records

SECONDARY OUTCOMES:
Prevalence of medical diseases and geriatric syndromes | Through study completion, an average of one month.
  Clinical and demographical conditions, and geriatric syndromes

CONTACTS AND LOCATIONS:
Overall Officials: Murielle MS Surquin, MD PhD, Principal Investigator — CHU Brugmann, Director of the Geriatrics Department
Locations (1):
- CHU Brugmann, Brussels, Belgium

REFERENCES:
- [Background] Mendes A, Serratrice C, Herrmann FR, Genton L, Perivier S, Scheffler M, Fassier T, Huber P, Jacques MC, Prendki V, Roux X, Di Silvestro K, Trombert V, Harbarth S, Gold G, Graf CE, Zekry D. Predictors of In-Hospital Mortality in Older Patients With COVID-19: The COVIDAge Study. J Am Med Dir Assoc. 2020 Nov;21(11):1546-1554.e3. doi: 10.1016/j.jamda.2020.09.014. Epub 2020 Sep 15. PMID 33138936
- [Background] Menager P, Briere O, Gautier J, Riou J, Sacco G, Brangier A, Annweiler C, Geria-Covid Study Group OBOT. Regular Use of VKA Prior to COVID-19 Associated with Lower 7-Day Survival in Hospitalized Frail Elderly COVID-19 Patients: The GERIA-COVID Cohort Study. Nutrients. 2020 Dec 24;13(1):39. doi: 10.3390/nu13010039. PMID 33374341
- [Background] Miralles O, Sanchez-Rodriguez D, Marco E, Annweiler C, Baztan A, Betancor E, Cambra A, Cesari M, Fontecha BJ, Gasowski J, Gillain S, Hope S, Phillips K, Piotrowicz K, Piro N, Sacco G, Saporiti E, Surquin M, Vall-Llosera E. Unmet needs, health policies, and actions during the COVID-19 pandemic: a report from six European countries. Eur Geriatr Med. 2021 Feb;12(1):193-204. doi: 10.1007/s41999-020-00415-x. Epub 2020 Oct 15. PMID 33057981